CLINICAL TRIAL: NCT02006862
Title: Olanzapine in Standard Clinical Practice. 6-month Efficacy and Safety Monitoring
Brief Title: eVAluatIon of OLanzapine TreatmEnT
Acronym: VIOLET
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2013-OLZ-EL-40
Record Dates: First submitted 2013-12-02; First posted 2013-12-10 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2014-08

CONDITIONS: Bipolar Disorder; Schizophrenia
Keywords: olanzapine; olanzapine treatment efficacy
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- olanzapine, schizophrenia

SUMMARY:
This clinical observational study aims to investigate the efficacy of olanzapine (Villamos ®) in accordance with the instructions attached thereto in standard clinical practice, followed by the physician to the patient.

This is a multicenter, non- interventional observational study , 6-month period without preparing the patient to take the usual his medication . A total of 3 scheduled visits : Visit 1 to Day 0 ( integration , base ) , Visit 2 at month 3 and Visit 3 at month 6 ( = end of treatment) .

The purpose of the study is to demonstrate the efficacy and safety of olanzapine in patients who are indicated . Will be monitored and recorded all the different concomitant therapy . The treatment of each patient is an individual designated by the physician , according to standard clinical practice and without any intervention research purpose .

During the six months of observation patients visit the clinic at the beginning (day 0 ), intermediate ( 3 months ) and end (month 6). The purpose of these visits is regularly monitored by their doctor for senile dementia and their behavior .

DETAILED DESCRIPTION:
Schizophrenia

Treatment may be divided as follows :

Treating first episode- Treatment of acute- Maintenance therapy , relapse prevention - Treatment -resistant schizophrenia Treating first episode

• The oral antipsychotics ( APS ) second generation ( atypical ) considered the treatment of choice : olanzapine , risperidone , quetiapine , aripiprazole , ziprasidone , amisulpride , paliperidone

* Sertindole used in patients who can not tolerate at least one of the remaining APS
* Advantages monotherapy
* The dose of medication ( FA ) is preferable to the lower limits of normal dose as defined
* The appropriate duration of therapy should be continued for 12-24 months after the recession of the episode .

Treatment of acute phase .

* first-line treatment is oral second generation APS . The doses appropriate to move within the therapeutic range as defined
* For patients who received first-generation APS and had either reduced efficacy or intolerable side effects, the treatment of choice is to switch to oral second-generation APS
* If patients receiving first-generation APS with good response and no side effects , remain in these
* The length of acute treatment is six weeks less
* Where there is a risk of increased body weight ( BW) or onset of diabetes mellitus ( DM ) as the treatment with atypical APS requires close monitoring and control routine Investigations
* After the acute phase and high rates of relapse , treatment appropriate to continue for 12-24 months
* If it is determined appropriate treatment discontinuation should be done gradually and with close monitoring to identify relapse symptoms
* In cases of acute psychotic and / or stimulants patients is necessary rapidly quelled . In these cases, the oral preparations are to be preferred . If required injectable formulations , the drugs of choice is lorazepam , haloperidol , olanzapine , ziprasidone , aripiprazole intramuscular administration.
* In each case of using haloperidol appropriate be combined with anticholinergic . Is not necessary to monitor the vital signs of the patient.

Maintenance therapy , relapse prevention

* If the patient has benefits the acute phase of a particular FA continue the same
* For oral or injectable long-acting antipsychotic used in maintenance therapy
* For patients who received first-generation APS who had either reduced efficacy or intolerable side effects, the treatment of choice is to switch to oral second -generation APS
* If patients receiving first-generation APS with good response and no side effects , remain in these
* Where there is a risk of increased OR for diabetes or as to the treatment with atypical antipsychotics should be closely monitored and Investigations routine check or even switch to another atypical or typical APS
* If the patient is happy with a VAT does not modify
* We prefer monotherapy
* The duration of therapy appropriate to be extended by 5.2 years for patients with a relapse and more than five years (perhaps lifelong ) for more than one relapse
* If the patient has received at least two APS ( including one informal ) for at least 6-8 weeks each without adequate clinical response , consider the resistant form of the disease and the possibility of using clozapine . In some cases it is useful to add a second APS to treatment with clozapine
* Long-acting APS is an option for the treatment if the patient's wishes or when there are issues of adherence to treatment. The long acting formulations should be prescribed to a specified limit .

resistant schizophrenia

* Examine possible factors of non-response in FA : dose , duration, compliance , substance abuse , physical illness , polypharmacy
* If the disease is refractory to treatment with standard APS , the clinician may initially tried using informal APS
* If the patient has received at least two APS ( including one informal ) for at least 6-8 weeks each without adequate clinical response , consider the resistant form of the disease and the possibility of using clozapine as soon as possible
* In some cases it is useful to add a second APS to treatment with clozapine .

Bipolar I Disorder A. manic / hypomanic or mixed EPISODE Step 1 - the first choice therapy : lithium, valproate , atypical antipsychotics ( aripiprazole, ziprasidone , quetiapine , olanzapine, risperidone ) , lithium or valproate + atypical antipsychotics ( aripiprazole, ziprasidone , quetiapine , olanzapine, risperidone ) with or without a benzodiazepine ( lorazepam ) at severe mania

* Necessary discontinuation of antidepressants.
* When selecting the first choice drug taken into account the personal and family history of response to treatment , tolerance , contraindications , drug interactions , comorbid conditions , symptoms of mania ( euphoric , dysphoric , psychotic ) and cost.

Step 2 (for inadequate response after 2 weeks) :

Optimizing a dose control in plasma levels , compliance check b Change to another drug first choice c Add another drug first choice

Step 3 (for inadequate response after an additional 2-4 weeks ) :

a change to another drug first choice b Start the second treatment option :

* Conventional antipsychotics ( haloperidol , chlorpromazine )
* Other atypical antipsychotics ( clozapine , paliperidone )
* Lithium or valproate + haloperidol
* carbamazepine
* Lithium + valproate , lithium + carbamazepine
* Electroconvulsive

Resistant cases:

- Add or change amisulpride , nimodipine

Not recommended :

* Monotherapy with gabapentin , pregabalin , topiramate , lamotrigine , tiagabine , verapamil
* Risperidone or olanzapine + carbamazepine

  * Recommended treatment continued for at least 6-12 months after remission .
  * Strong dose reduction after the recession as tolerated . B. Depressive Episode

Step 1 - Cure first choice :

* Lithium , lamotrigine , quetiapine
* Lithium or divalproex + SSRI or bupropion, olanzapine + SSRI, lithium + valproate

  * When selecting the first choice drug taken into account the personal and family history of response to treatment , tolerance , contraindications , drug interactions , comorbid conditions, severity of depression, suicidality , and cost.
  * Antidepressants , when granted , should always be combined with antimanic agent ( lithium, valproate , atypical antipsychotic )
  * When coexisting psychotic symptoms should be added and atypical antipsychotic .

Step 2 ( inadequate response after 4 weeks) :

Optimizing a dose control in plasma levels , compliance check b Add or change to another treatment first choice

Step 3 ( inadequate response after 4 weeks) :

a change to another drug first choice b Start the second treatment option :

* Quetiapine + SSRI
* Valproate , lithium or valproate + lamotrigine

Step 4 - Treatment option 3 ( inadequate response after 4 weeks) :

* Carbamazepine , lithium + carbamazepine
* Olanzapine
* Lithium or valproate + venlafaxine or mirtazapine , lithium or valproate or atypical antipsychotic + tricyclic antidepressant , lithium + MAO inhibitor
* Lithium or valproate or carbamazepine + SSRI + lamotrigine
* Electroconvulsive therapy : particularly in patients with severe stroke, accompanying psychotic or catatonic symptoms , high risk of suicidality , refusing to take food , pregnancy may be the first choice

Not recommended :

* Monotherapy with gabapentin
* Monotherapy with aripiprazole

  * Recommended maintenance antidepressant to 12 weeks and then gradually discontinued within four weeks unless diversion occurs in mania or hypomania earlier.

CAUTION - MAINTENANCE

Treatment first choice :

* Lithium (if probable good compliance in the future) , valproate ( avoided in women of childbearing age ) , lamotrigine
* Aripiprazole, quetiapine , olanzapine , risperidone or risperidone depot
* Lithium or valproate + quetiapine adjunctive treatment with risperidone or risperidone depot, additional treatment with ziprasidone • Start after a severe manic episode or after two episodes ( manic , mixed or depressive )

  * When selecting the first choice drug taken into account the personal and family history of response to treatment , tolerance , contraindications , drug interactions , gender , comorbid conditions, compliance history , the prevalence of manic or depressive symptoms and costs.
  * a) When prevailing manic / hypomanic episodes : lithium, valproate , aripiprazole , quetiapine , olanzapine monotherapy or combinations b ) When the prevailing depressive episodes quetiapine or lamotrigine antimanic + ( + antidepressant in a limited number of patients )

Treatment 2nd choice :

* carbamazepine
* Lithium + valproate , lithium + carbamazepine , lamotrigine , lithium +
* Lithium or divalproex + olanzapine , lithium + risperidone , olanzapine + fluoxetine

Treatment option 3 :

- Adjunctive therapy with gabapentin

* Adjunctive therapy with clozapine
* Adjunctive therapy with omega- 3 fatty acids
* Additional maintenance electroconvulsive therapy

We recommended :

- Monotherapy : gabapentin , topiramate , antidepressants

* It is recommended continued treatment for at least 2 years after an episode of illness and up to 5 years if there are risk factors for relapse ( substance use , psychotic symptoms , history of frequent relapses , ongoing stressful life events , poor psychosocial support)
* Recommended continued treatment indefinitely if it is effective in preventing recurrence .

Anxiety & Related Disorders Generalised Anxiety Disorder

Step 1 - Cure first choice :

- The SSRIs escitalopram , paroxetine , sertraline or SNRIs venlafaxine, duloxetine with or without benzodiazepines ( alprazolam , diazepam to 2-4 weeks )- pregabalin

* Preferred antidepressants (SSRIs, SNRIs) when coexisting depression .
* When selecting the first choice drug taken into account the individual and family history of response to treatment , tolerance , contraindications , drug interactions , comorbid conditions , the risk of suicidality and costs.

Step 2 (for insufficient response after 8-12 weeks ) :

a dose increase b change to another drug first choice c addition or change to the second drug of choice :

* quetiapine
* Benzodiazepines ( alprazolam , diazepam ) when there is no history dependence
* hydroxyzine
* buspirone

Resistant cases:

* Add another atypical antipsychotic ( olanzapine , risperidone )
* Addition of valproate
* Addition of a beta-blocker ( control somatic symptoms) Recommended continued treatment for at least 6-12 months after response. Panic Disorder

Step 1 - Cure first choice :

* SSRIs ( escitalopram , paroxetine , sertraline , citalopram , fluvoxamine , fluoxetine) or venlafaxine with or without benzodiazepines ( alprazolam , diazepam , lorazepam to 2-4 weeks )
* Monotherapy with benzodiazepines for 2-4 weeks when not coexist depressive symptoms • When selecting the first choice drug taken into account the individual and family history of response to treatment , tolerance , contraindications , the drug interactions , comorbid conditions , risk suicidality and costs.

Step 2 (for insufficient response after 8-12 weeks ) :

a dose increase b change to another drug first choice c Treatments second choice :

* Switch to clomipramine
* Addition of benzodiazepines ( alprazolam , diazepam , lorazepam ) for longer periods of time when there is no history dependence

Resistant cases:

* Combination of drugs first or second choice ( eg clomipramine or SSRI + venlafaxine )
* Addition of atypical antipsychotic
* Addition of valproate or lithium
* Addition or change to mirtazapine
* Change in moclobemide Recommended continued treatment at the same dose for at least 12-24 months after response . Social Anxiety Disorder ( Social Phobia )

Step 1 - Cure first choice :

- SSRIs ( escitalopram , paroxetine , sertraline , citalopram , fluvoxamine , fluoxetine) or venlafaxine with or without benzodiazepines ( bromazepam , clonazepam to 2-4 weeks)

* When selecting the first choice drug taken into account the individual and family history of response to treatment , tolerance , contraindications , the drug interactions , comorbid conditions , risk suicidality and costs.

Step 2 (for insufficient response after 8-12 weeks ) :

a dose increase b change to another drug first choice c Treatments second choice :

* Change in moclobemide
* Addition of a benzodiazepine ( clonazepam ) for longer periods of time when there is no history dependence

Resistant cases:

* The first choice drug combination ( eg SSRI + venlafaxine )
* Addition of atypical antipsychotic ( olanzapine )
* Addition of pregabalin
* Addition or change to mirtazapine
* Addition of buspirone Recommended continued treatment at the same dose for at least 6-12 months after response . obsessive Compulsive Disorder Step 1 - Cure first choice : - SSRIs ( escitalopram , paroxetine , sertraline , citalopram , fluvoxamine , fluoxetine) with titration to the maximum tolerated dose

  * usually needed higher doses than for addressing depression or other anxiety disorders .
  * When selecting the first choice drug taken into account the individual and family history of response to treatment , tolerance , contraindications , drug interactions , comorbid conditions , the risk of suicidality and costs.

Step 2 (for inadequate response after 8 to 12 weeks, of which at least 4-6 weeks at the maximum tolerated dose) : a change to another drug first choice b switch to clomipramine (2nd choice )

Resistant cases:

* Addition of haloperidol or atypical antipsychotic ( aripiprazole , quetiapine , olanzapine , risperidone )
* Combination of SSRI + clomipramine
* Addition or change to venlafaxine, mirtazapine
* Addition of lithium
* Addition of buspirone Recommended continued treatment at the same dose for at least 12-24 months after response . Post Traumatic Stress Disorder

  1. st choice : paroxetine , sertraline , fluoxetine or venlafaxine

     • When selecting the first choice drug taken into account the individual and family history of response to treatment , tolerance , contraindications , drug interactions , comorbid conditions and costs.
  2. nd choice :
* amitriptyline
* mirtazapine
* lamotrigine
* risperidone

Option 3 :

* Citalopram , escitalopram , fluvoxamine , moclobemide
* Olanzapine , quetiapine
* carbamazepine

Resistant cases:

* A combination of the first or second drug of choice
* Addition of olanzapine , risperidone , quetiapine Recommended continued treatment at the same dose for at least 6-12 months after response .

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and over

  * Diagnosis of schizophrenia (DSM-IV-DR)
  * Maintaining the clinical improvement during continuation therapy in patients who have shown an initial treatment response .
  * Treatment of moderate to severe manic episode .
  * Patients whose manic episode has responded to olanzapine treatment ,
  * for the prevention of recurrence in patients with bipolar disorder (DSM-IV-)
  * The patient has a reliable caregiver
  * Signed consent form to participate in the study after informed by reliable caregiver of the patient or other witness
  * The patient is treated with olanzapine before joining the present study
  * The patient had conformability to study

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the ingredients.

  * Patients with known risk for narrow-angle glaucoma .
  * Dementia-related psychosis and / or behavioral disturbances
  * Disease Parkinson
  * Neuroleptic Malignant Syndrome (NMS)
  * Patients with low leukocyte and / or neutrophil counts for any reason, in patients receiving medicines known to cause neutropenia ,
  * Clinically significant laboratory and ECG abnormalities .
  * Participation in another clinical study than this
  * Refusal to sign the consent form to participate in the study after informed by reliable caregiver of the patient or other witness
  * The patient is treated with olanzapine before joining the clinical trial

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with schizophrenia or bipolar disorders
Sampling Method: Non-Probability Sample
Enrollment: 468 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in scales' ratings to assess efficacy | baseline, 3 months, 6 months
  change in PANSS rating change in Y-MRS rating change in CES-D rating

SECONDARY OUTCOMES:
Safety assessment | baseline, 3 months, 6 months
  Number of Adverse Events - Serious Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Agia Olga Konstantopouleion Hospital, Athens, Greece